CLINICAL TRIAL: NCT05581394
Title: Accuracy of BabySat V3 With Profound Hypoxia and Motion
Status: Completed | Type: Observational
Sponsor: Owlet Baby Care, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: BICK-ACC-20220714
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BabySat V3 — Evaluation of Accuracy of BabySat V3

SUMMARY:
Performance testing of pulse oximeters. The protocol involves brief stable arterial oxygen desaturation in healthy volunteers and sampling arterial blood when a stable level of hypoxia has been attained and during different motion scenarios. The blood sample is analyzed for oxygen saturation with a gold standard bench CO-oximeter. This protocol is aligned with the latest ISO and FDA guidance documents for pulse oximeter testing.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, aged ≥18 and <50
* The subject is in good general health with no evidence of any medical problems
* The subject is fluent in both written and spoken English
* The subject has provided informed consent and is willing to comply with the study procedures

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in this study should be healthy, between 18 and 50 years of age and willing to participate in breathing studies with blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of accuracy during motion | During the oxygen desaturation assessment
  Determine the accuracy during varying degrees of motion and oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: John Feiner, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University California San Fransisco, Department of Anesthesia, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No